CLINICAL TRIAL: NCT03805698
Title: Use of Platelet Rich Plasma After Arthroscopic Debridement for Triangular Fibrocartilage Complex Tears
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID stopped surgeries
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, David Kulber, MD, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00053449
Record Dates: First submitted 2019-01-07; First posted 2019-01-16 (Actual); Results first posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Arthroscopic Surgery; Triangular Fibrocartilage Complex Injury
Keywords: Platelet-rich Plasma
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patients undergoing arthroscopic debridement for triangular fibrocartilage complex (TFCC) tears will be treated with PRP (24 subjects) versus no treatment with Platelet-rich plasma (PRP) (24 subjects).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Platelet-rich Plasma (PRP) group (Experimental): Twenty-four (24) subjects undergoing arthroscopic debridement for triangular fibrocartilage complex (TFCC) tears will be treated intraoperatively with platelet-rich plasma (PRP) (24 subjects).
  Intervention: use of Cascade device; Autologous Fibrin & Platelet System; once processed, the platelet-rich plasma (PRP)is injected into the debrided wrist
  Interventions: Device: Platelet-rich Plasma (PRP)
- Standard Treatment group (Active Comparator): Twenty-four (24) subjects undergoing arthroscopic debridement for triangular fibrocartilage complex (TFCC) tears will undergo treatment, as is standard of care, followed by no treatment with platelet-rich plasma (PRP)(24 subjects).
  Intervention: No platelet-rich plasma (PRP) injection into debrided wrist
  Interventions: Other: Standard Arthroscopic Debridement

INTERVENTIONS:
Device: Platelet-rich Plasma (PRP) — The CASCADE Autologous Platelet System is a product made commercially available by the Musculoskeletal Transplant Foundation (MTF) for PRP processing. Once processed, the PRP is injected into the debrided wrist.
  Other Names: PRP group; Treatment group
  Arms: Platelet-rich Plasma (PRP) group
Other: Standard Arthroscopic Debridement — Standard arthroscopic debridement. No PRP injection.
  Other Names: Standard Treatment; Control group
  Arms: Standard Treatment group

SUMMARY:
The objective of this study is to compare outcomes and functionality measures of subjects treated with platelet rich plasma (PRP) after arthroscopic debridement of triangular fibrocartilage complex (TFCC) tears to subjects treated with arthroscopic debridement alone.

DETAILED DESCRIPTION:
Patients with triangular fibrocartilage complex (TFCC) tears will undergo treatment with arthroscopic debridement, as is standard of care, followed by treatment with platelet rich plasma (PRP) (24 subjects) versus no treatment with PRP (24 subjects). Outcome measures will include Modified Mayo Wrist scores (pain scale scores, grip strength, wrist range of motion, functional status) and Patient-rated Wrist Evaluation (PRWE) scores.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female >18 years of age
* triangular fibrocartilage complex (TFCC) tear requiring surgical intervention
* Be willing to undergo arthroscopic debridement and injection with platelet-rich plasma (PRP)
* Be in good health other than the TFCC tear
* Have realistic expectations of surgical results
* Understand and be willing to follow all aspects of the study protocol and have signed and dated the IRB-approved Informed Consent Form and the Authorization for Use and Release of Health and Research Study Information (HIPAA) form prior to any study-related procedures being performed

Exclusion Criteria:

* Have collagen-vascular, connective tissue, or bleeding disorders
* Be a smoker or have smoked in last 2 months
* Have any disease, including uncontrolled diabetes, which is clinically known to impact wound healing ability
* Have regional sympathetic dystrophy
* Be pregnant, lactating or expecting to be within the next 24 months
* Currently have an alcohol/substance abuse problem or have had a relapse within one year to screening visit
* Have an abscess or infection at the time of surgery
* Have a condition or be in a situation that, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kulber, MD, Principal Investigator — Cedars-Sinai
Locations (1):
- Cedars-Sinai Department of Hand Surgery, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: medical clinic from 07/22/19-02/02/2020
Groups:
- Platelet-rich Plasma (PRP) Group: Twenty-four (24) subjects undergoing arthroscopic debridement for TFCC tears will be treated intraoperatively with PRP (24 subjects).
  Intervention: use of Cascade device; Autologous Fibrin & Platelet System; once processed, the PRP is injected into the debrided wrist
  Platelet-rich Plasma (PRP): The CASCADE Autologous Platelet System is a product made commercially available by the Musculoskeletal Transplant Foundation (MTF) for PRP processing. Once processed, the PRP is injected into the debrided wrist.
- Standard Treatment Group: Twenty-four (24) subjects undergoing arthroscopic debridement for TFCC tears will undergo treatement, as is standard of care, followed by no treatment with PRP (24 subjects).
  Intervention: No PRP injection into debrided wrist
  Standard Arthroscopic Debridement: Standard arthroscopic debridement. No PRP injection.
Period: Overall Study
Arm/Group | Platelet-rich Plasma (PRP) Group | Standard Treatment Group
Started | 10 | 0
Completed | 10 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: study not completed due to COVID shutdown
Groups:
- Total: Total of all reporting groups
Arm/Group | Platelet-rich Plasma (PRP) Group | Standard Treatment Group | Total
Number analyzed (Participants) | 10 | 0 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 9 |  | 9
  >=65 years | 1 |  | 1
Age, Continuous [Mean (Full Range); unit: years] | 54.9 [30 to 76] |  | 54.9 [30 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 |  | 7
  Male | 3 |  | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 |  | 10

OUTCOME MEASURES:

1. Primary Outcome: Patient-rated Wrist Evaluation (PRWE) Scores
Description: The Patient-rated Wrist Evaluation is a 15 item patient-reported questionnaire to assess change from pre to post-op that asks the patient to rate their pain and function on a 10-point scale. 0 (minimum) means no pain/did not experience functional difficulties and 10 (maximum) means the worst pain/difficulty to function. Total minimum is 0 and total maximum for this scale measure is 150.
  Compare Mean patient-rated Wrist Evaluation outcome scores from pre-op to post-op.
Time Frame: change from pre to post-op
Population: The intervention was incomplete due to COVID and questionnaires were not obtained.
Arm/Group | Platelet-rich Plasma (PRP) Group | Standard Treatment Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Modified Mayo Wrist Score - Grip Strength Score
Description: Modified Mayo Wrist score - Grip strength score: A change in grip strength from pre to post-op (percentage of normal) - on 0 (minimum/total)-100% (maximum/total) scale between patients treated with PRP vs. patients not treated with PRP after arthroscopic debridement.
  Compare mean (percentage of normal) Grip strength scores from pre-op to post-op.
Time Frame: Up to 5 time points (change from pre to post-op): pre-op, post op: month 1, month 3, month 6 and year 1; Subjects will be followed for 12 months post arthroscopic debridement.
Population: The Grip strength score was not obtained.
Arm/Group | Platelet-rich Plasma (PRP) Group | Standard Treatment Group
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Modified Mayo Wrist Score - Pain Score
Description: Modified Mayo Wrist score - Mean Pain score change assessment from pre to post-op: 0 (minimum/total; severe to intolerable)-25 (maximum/total; no pain) point scale
Time Frame: Up to 5 time points (change from pre to post-op): pre-op, post op: month 1, month 3, month 6 and year 1
Population: Measurement was not obtained for any subject.
Arm/Group | Platelet-rich Plasma (PRP) Group | Standard Treatment Group
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Modified Mayo Wrist Score - Range of Motion Score
Description: Modified Mayo Wrist score - Range of motion score: Assessment of change from pre to post-op in patient's range of motion (percentage of normal) on a 0 (minimum/total)-100% (maximum/total) scale between mean patient score of patients treated with PRP vs. patients not treated with PRP after arthroscopic debridement.
Time Frame: as for outcome 2
Population: The wrist score was not obtained for any patient in the study.
Arm/Group | Platelet-rich Plasma (PRP) Group | Standard Treatment Group
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Modified Mayo Wrist Score - Functional Status Score
Description: Modified Mayo Wrist score - Functional status score: An assessment to review mean change from pre to post-op) 0 (minimum)-25 (maximum) point scale; a score of 0 denotes patient's inability to work because of pain and 25 denotes patients ability to work/return to regular employment
Time Frame: as for outcome 2
Population: Wrist score was not obtained for any subject.
Arm/Group | Platelet-rich Plasma (PRP) Group | Standard Treatment Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: no additional adverse event collected
Groups:
- Platelet-rich Plasma (PRP) Group: Twenty-four (24) subjects undergoing arthroscopic debridement for triangular fibrocartilage complex (TFCC) tears will be treated intraoperatively with Platelet-rich Plasma (PRP) (24 subjects).
  Intervention: use of Cascade device; Autologous Fibrin & Platelet System; once processed, the PRP is injected into the debrided wrist
  Platelet-rich Plasma (PRP): The CASCADE Autologous Platelet System is a product made commercially available by the Musculoskeletal Transplant Foundation (MTF) for Platelet-rich Plasma (PRP) processing. Once processed, the Platelet-rich Plasma (PRP) is injected into the debrided wrist.
- Standard Treatment Group: Twenty-four (24) subjects undergoing arthroscopic debridement for triangular fibrocartilage complex (TFCC) tears will undergo treatment, as is standard of care, followed by no treatment with Platelet-rich Plasma (PRP) (24 subjects).
  Intervention: No Platelet-rich Plasma (PRP) injection into debrided wrist
  Standard Arthroscopic Debridement: Standard arthroscopic debridement. No Platelet-rich Plasma (PRP) injection.
Arm/Group | Platelet-rich Plasma (PRP) Group | Standard Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/0
Other Adverse Events (participants affected / at risk) | 0/10 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT03805698/Prot_SAP_003.pdf
  • Informed Consent Form (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT03805698/ICF_004.pdf